CLINICAL TRIAL: NCT04317079
Title: Evaluation of the Effects of the Administration of 5 Milligrams and 15 Milligrams of Hydroxytyrosol, an Extra Virgin Olive Oil Phenolic Compound, Versus Placebo, Combined With Diet, in Anthropometric Parameters in Overweight and Obese Women
Brief Title: Effects of Hydroxytyrosol Administration in Anthropometric Parameters in Overweight and Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Alexandros Kokkinos, Associate Professor in Internal Medicine, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HydroxytyrosolStudy
Record Dates: First submitted 2020-03-19; First posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Body Weight; Visceral Obesity
Keywords: Hydroxytyrosol; Body weight; Visceral fat
MeSH Terms: conditions — Body Weight; Obesity, Abdominal | interventions — 3,4-dihydroxyphenylethanol; Diet

STUDY DESIGN:
Intervention Model Description: Administration of hydroxytyrosol (15mg versus 5 mg daily) versus placebo for 6 months in combination with diet in order to assess effects in body weight, body fat mass and visceral fat mass loss
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 15mg of hydroxytyrosol (Active Comparator): 15 milligrams of hydroxytyrosol given as 2 capsules containing 2.5mg of hydroxytyrosol each given three times daily before main meals (totally 6 capsules daily) in combination with diet
  Interventions: Dietary Supplement: Hydroxytyrosol; Other: Diet
- 5mg of hydroxytyrosol (Active Comparator): 5 milligrams of hydroxytyrosol given as 2 capsules containing 2.5mg of hydroxytyrosol each given in the morning and at night before meals and 2 capsules of placebo before lunch (totally 6 capsules daily) in combination with diet
  Interventions: Dietary Supplement: Hydroxytyrosol; Other: Diet
- placebo (Placebo Comparator): 2 capsules of placebo given 3 times daily before meals (totally 6 capsules daily) in combination with diet
  Interventions: Other: Diet

INTERVENTIONS:
Dietary Supplement: Hydroxytyrosol — Administration of hydroxytyrosol in doses 15mg and 5 mg compared to placebo for 6 months
  Arms: 15mg of hydroxytyrosol; 5mg of hydroxytyrosol
Other: Diet — Consultation by a dietitian was offered to all participants

SUMMARY:
This study aims to investigate the potential effects of the administration of hydroxytyrosol, which is an extra virgin olive oil phenolic compound, in doses 15 milligrams and 5 milligrams daily versus placebo for 6 months in anthropometric parameters such as body weight, body fat and visceral fat, in combination with diet, in overweight and obese women.

DETAILED DESCRIPTION:
Hydroxytyrosol is an extra virgin olive oil phenolic compound which has known protective effects in LDL oxidation and reduces oxidative stress. Olive oil has been associated with enhanced weight loss, and hydroxytyrosol could have a potential role in this.

Participants entered the study after signing the informed consent document. Detailed medical and family history was taken at baseline visit, and measurement of height, body weight, body fat and visceral fat were also made. Each participant visited a dietitian the same day and written consultation concerning the diet to be followed was given, based on Mediterranean diet and 500 kilocalories below their estimated Basal Metabolic Rate. The above measurements and dietitian consultation were repeated in each visit during the intervention (4,12 and 24 weeks).

Baseline laboratory testing was made including urea, creatinine, aminotransferases and fasting lipids and glucose, while serum and plasma were stored in -80 Celsius degrees for future analyses. Blood samples were also taken at 4, 12 and 24 weeks of the intervention.

All participants had an identical meal test at baseline, at 12 and 24 months and blood samples were collected at times 0, 30, 60, 90, 120, 150 and 180 minutes after meal consumption. Samples were also stored in -80 Celsius degrees for future analyses.

Each participant received in each visit prepackaged the quantity of capsules until the next scheduled visit, and the used empty blisters were returned in the following visit in order to assess compliance in capsules consumption. 24-hour diet recalls were used to assess compliance to diet.

In each visit an investigation concerning potential adverse events was made and data were recorded.

A communication was obtained with each participant who discontinued the study before 24 weeks, the reasons for discontinuation were recorded and data obtained until their last visit before study discontinuation were used in analyses.

Paired analyses were made using the system Statistical Package for the Social Sciences comparing all study groups before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

Overweight and obese women. Stable body weight (<5% variation) during the past 3 months before enrollment. Stable hypolipidemic treatment for at least 3 months before enrollment.

Exclusion Criteria:

* Diabetes mellitus
* Neoplasms
* Autoimmune conditions
* Psychiatric disorders (excluding stable depressive disorder)
* Hyper/hypo-thyroidism with recent changes in medical treatment during the past 6 months before enrollment
* Renal impairment, defined as estimated Glomerular Filtration Rate (MDRD) <60millilitres/min
* Heart failure, defined as left ventricle Ejection Fraction <40%, use of diuretics or other treatment due to heart failure (antihypertensive medications allowed)
* Impaired liver function, defined as liver transaminases values twice above the upper normal range
* Malabsorption status (inflammatory bowel disease, previous bariatric surgery, chronic pancreatitis)
* Medical treatment known to influence body weight (steroids, oestrogens/ progesterone, topiramate, mirtazapine or anti-obesity treatment)
* Unwillingness to participate to the study
* Baseline waist circumference >130cm due to technical difficulties in visceral fat measurement
* Pregnancy, lactation

Ages: 18 Years to 66 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Baseline, 4,12 and 24 weeks
  Measurement of body weight via TANITA Bioelectrical Impedance Analysis technology
Change in body fat mass | Baseline, 4,12 and 24 weeks
  Measurement of body fat mass via bioelectrical impedance (TANITA Bioelectrical Impedance Analysis technology)
Change in visceral fat | Baseline, 4, 12 and 24 weeks
  Measurement via TANITA technology

SECONDARY OUTCOMES:
Changes in blood lipids | Baseline, 12 and 24 weeks
  Measurement of serum total cholesterol, high-density lipoprotein and triglycerides
Changes in blood glucose | Baseline, 12 and 24 weeks
  Measurement of serum glucose
Changes in blood insulin | Baseline, 12 and 24 weeks
  Measurement of serum insulin

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Tentolouris, MD,PhD, Principal Investigator — National Kapodistrian University of Athens
Locations (1):
- Diabetes Clinical Research Laboratory, 1st Department of Propaedeutic Internal Medicine, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cotrim BA, Joglar J, Rojas MJ, del Olmo JM, Macias-Gonzalez M, Cuevas MR, Fito M, Munoz-Aguayo D, Planells MI, Farre M, de Fonseca FR, de la Torre R. Unsaturated fatty alcohol derivatives of olive oil phenolic compounds with potential low-density lipoprotein (LDL) antioxidant and antiobesity properties. J Agric Food Chem. 2012 Feb 1;60(4):1067-74. doi: 10.1021/jf203814r. Epub 2012 Jan 20. PMID 22220510
- [Background] Peyrol J, Riva C, Amiot MJ. Hydroxytyrosol in the Prevention of the Metabolic Syndrome and Related Disorders. Nutrients. 2017 Mar 20;9(3):306. doi: 10.3390/nu9030306. PMID 28335507
- [Background] Colica C, Di Renzo L, Trombetta D, Smeriglio A, Bernardini S, Cioccoloni G, Costa de Miranda R, Gualtieri P, Sinibaldi Salimei P, De Lorenzo A. Antioxidant Effects of a Hydroxytyrosol-Based Pharmaceutical Formulation on Body Composition, Metabolic State, and Gene Expression: A Randomized Double-Blinded, Placebo-Controlled Crossover Trial. Oxid Med Cell Longev. 2017;2017:2473495. doi: 10.1155/2017/2473495. Epub 2017 Aug 9. PMID 28855976